CLINICAL TRIAL: NCT05684783
Title: Developing the Role of Dementia Champions in the Homecare Sector
Brief Title: Dementia Champions in Homecare
Acronym: DemChamp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 320561
Record Dates: First submitted 2022-12-13; First posted 2023-01-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-12

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 interviews: Care professionals with experience of being or working with Dementia Champions, and people affected by dementia who have received care from services with Dementia Champions.
- Group 2 interviews: Homecare professionals working in services where there are no Dementia Champions, and people affected by dementia who have received care from services with no Dementia Champions.

SUMMARY:
This is a descriptive, explorative study in which we will explore how the role of Dementia Champions in homecare services could develop, and become more widely implemented in this sector's workforce.

DETAILED DESCRIPTION:
This study had three parts:

1. The investigators will start by learning from the work of other Dementia Champions working across care services to get a 'real world' in-depth understanding of what working as a Dementia Champion involves, what works well, and what can be improved. The investigators will carry out qualitative interviews with care professionals with experience of being or working with Dementia Champions. They will also speak to people affected by dementia (people living with dementia and their family carers) who have received care from services with Dementia Champions.
2. The investigators will carry out a stakeholder consultation workshop with 10 people including care professionals, people affected by dementia, and other relevant stakeholders, to build on what we have learned so far. They will commission a Science Illustrator to visually scribe the workshop discussions and produce an illustration of the Dementia Champion in homecare role.
3. The investigators will use the model created in part 2 of the study to facilitate interviews in part 3. They will speak to staff working in homecare services (managers and homecare workers) that do not have Dementia Champions in them, and people living with dementia and family members who use homecare services that do not have Dementia Champions in them. This will help the research team understand how to better establish the role of Dementia Champions and how this could work within homecare, including what would be needed to support staff in this role.

ELIGIBILITY:
Inclusion criteria

Part 1 (group 1 interviews):

* Staff who are or have been DCs in services that provide care and support to people affected by dementia
* Staff who work or have worked alongside DCs in services that provide care and support to people affected by dementia
* Staff with expertise in dementia e.g. those from third sector or voluntary dementia organisations
* A person living with dementia who receives or has received support or care from services with DCs embedded within the team i.e., homecare
* A current or former family carer of a person living with dementia who receives or has received support or care from services with DCs embedded within the team i.e., homecare

Part 2 (stakeholder consultation workshop):

* Homecare staff (including any DCs identified from previous study phases)
* Dementia specialists (e.g., social workers with expertise in dementia, Admiral Nurses)
* People living with dementia in receipt of homecare support
* Current or former family carers of a person living with dementia in receipt of homecare support
* Any other relevant care staff

Part 3 (group 2 interviews):

* A homecare worker, manager, or other member of homecare staff
* A person living with dementia in receipt of homecare support
* A current or former family carer of a person living with dementia in receipt of homecare

Exclusion Criteria:

* People who do not have capacity to consent to take part in this research study. The research team has experience of conducting informal assessments of capacity, using the three-stage test outlined in the Mental Capacity Act 2005 of England and Wales.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants from England, Scotland, Wales, or Northern Ireland who either, recruited from health or social care settings.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
This is a qualitative study involving interviews and as such, there are no measurable outcomes. We will, however, use an interview topic guide to conduct interviews, and use the findings to produce a Model of Dementia Champions in the homecare sector | 8 months
  Experiences of care staff, people living with dementia, and family carers of dementia champions in homecare.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Leverton, Principal Investigator — King's College London
Locations (1):
- Home Instead Devon, South Molton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
If participants agree to their interview data being used for future ethically approved research by King's College London then we will make this available to other King's College London researchers.